CLINICAL TRIAL: NCT03150511
Title: Tesamorelin Therapy to Enhance Axonal Regeneration, Minimize Muscle Atrophy, and Improve Functional Outcomes Following Peripheral Nerve Injury
Brief Title: Tesamorelin to Improve Functional Outcomes After Peripheral Nerve Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00110936-2; W81XWH-16-C-0188 (Other Grant/Funding Number: Department of Defense); W81XWH-22-1-0257 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2017-04-19; First posted 2017-05-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — tesamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tesamorelin treatment (Experimental)
  Interventions: Drug: Tesamorelin 2 Milligrams (MG)
- No Drug (No Intervention)

INTERVENTIONS:
Drug: Tesamorelin 2 Milligrams (MG) — Daily self-administered study drug
  Other Names: Egrifta
  Arms: Tesamorelin treatment

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy of tesamorelin as a therapy for peripheral nerve injuries. The investigators hypothesize that treatment with tesamorelin will result in faster and more substantial recovery of motor and sensory function following surgical repair of injured peripheral nerves. Patients with upper extremity nerve injuries will be randomly assigned to receive either tesamorelin treatment or no treatment. Assessments for nerve regeneration, muscle function, and sensation will be conducted every three months for a total of 12 months. Outcomes in patients receiving tesamorelin will be compared to those in the untreated group to determine the effectiveness of tesamorelin as a therapeutic intervention for nerve injuries.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, clinical trial assessing the efficacy of tesamorelin as a therapy to improve functional recovery following peripheral nerve injury. Tesamorelin is a drug that stimulates increased production of growth hormone, and growth hormone has been shown to improve nerve regeneration and functional recovery in animal studies.

A total of 36 participants with repaired ulnar nerve lacerations will be enrolled, of which 18 will be randomly assigned to receive the study drug and 18 will receive no treatment. To minimize bias, outcome assessors and the biostatistician analyzing the data will be blinded to the treatment assignments. Following enrollment, each participant will have 12 monthly follow-up visits during which participants will undergo testing to assess recovery. Outcome assessments will include clinical exams, electrodiagnostic studies and questionnaires.

The total duration of the study is expected to be 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Ulnar nerve laceration at the wrist, repaired primarily

Exclusion Criteria:

* Certain cancers (active or in the past)
* Uncontrolled diabetes or hypertension
* Certain pituitary problems
* Oral contraceptives
* Pregnancy
* Drug or alcohol dependence
* Psychosocial issues that would limit participation and compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
3-point chuck pinch test | 12 months
  Pinch strength measure as measured by a pinch gauge.

SECONDARY OUTCOMES:
Disability of the Arm, Shoulder, and Hand (DASH) score | 12 months
  Questionnaire
Michigan Hand Questionnaire score | 12 months
  Questionnaire
Amplitude of response | 12 months
  Nerve conduction study measure
Latency of response | 12 months
  Nerve conduction study measure
Velocity of response | 12 months
  Nerve conduction study measure
Modified British Medical Research Council (MBMRC) sensory grading (S0-S4) | 12 months
  Standardized clinical assessment of sensory function using 2-point discrimination and monofilament testing. S0 indicates no recovery and S4 indicates full recovery.
Modified British Medical Research Council (MBMRC) motor grading (M0-M5) | 12 months
  Standardized clinical assessment of motor function. M0 indicates no muscle contraction and M5 indicates active range of motion against strong resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Sami Tuffaha, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sami Tuffaha, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No